CLINICAL TRIAL: NCT03582410
Title: Absorbable vs Non-absorbable Suture in Laparoscopic Sacral Colpopexy: a Randomized Controlled Trial
Brief Title: Different Types of Suture for Sacral Colpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Maurizio Guido, Clinical Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ospedale regionale F. Miulli
Record Dates: First submitted 2018-06-06; First posted 2018-07-11 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable suture (Active Comparator): laparoscopic sacral colpopexy with absorbable suture
  Interventions: Procedure: laparoscopic sacral colpopexy with absorbable suture
- Non absorbable suture (Active Comparator): laparoscopic sacral colpopexy with non absorbable suture
  Interventions: Procedure: laparoscopic sacral colpopexy with non absorbable suture

INTERVENTIONS:
Procedure: laparoscopic sacral colpopexy with absorbable suture — laparoscopic sacral colpopexy to correct pelvic organ prolapse with anterior and posterior meshes with absorbable suture
  Arms: Absorbable suture
Procedure: laparoscopic sacral colpopexy with non absorbable suture — laparoscopic sacral colpopexy to correct pelvic organ prolapse with anterior and posterior meshes with non absorbable suture
  Arms: Non absorbable suture

SUMMARY:
This randomized controlled study is designed to test absorbable suture compared to non absorbable suture in laparoscopic sacral colpopexy in terms of anatomical correction of the prolapse, post-operative and long term morbidity, rate of recurrence, subjective satisfaction of the patient and rate of mesh erosion.

ELIGIBILITY:
Inclusion Criteria:

* patients who required surgical treatment for symptomatic pelvic organ prolapse stage ≥ 2 with or without stress urinary incontinence

Exclusion Criteria:

* Age > 75 years
* Severe cardiovascular or respiratory disease
* Pregnancy

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with anatomical correction of the prolapse | 1 year
  Anatomical correction of the prolapse evaluated by gynecological visit

SECONDARY OUTCOMES:
rate mesh erosion | 1 year
long term outcomes | 1 year
  development of nicturia, dysuria, obstructed defecation , urinary incontinence
Rate of recurrence | 1 year
  de novo anterior or central or posterior compartment prolapse

CONTACTS AND LOCATIONS:
Locations (1):
- ospedale regionale Miulli, Acquaviva delle Fonti, Bari, Italy